CLINICAL TRIAL: NCT06512220
Title: Imaging the Effects of Serotonin 2A Receptor Modulation on Synaptic Density in Treatment-resistant Depression (SYNVEST)
Acronym: SYNVEST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Ishrat Husain, Senior Scientist, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 052-2022
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Treatment Resistant Depression
Keywords: Psilocybin; Psychedelics; Clinical Trial; Positron-Emission Tomography; Treatment Resistant Depression; Neurophysiology Testing
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risperidone (1 mg) + Psilocybin (25 mg) (Experimental): o One capsule of risperidone 1 mg will be taken first followed 60 minutes later by one capsule of psilocybin 25 mg. Both capsules will be taken orally with a glass of water.
  Interventions: Drug: Psilocybin 25 mg; Drug: Risperidone 1 MG
- Psilocybin (25 mg) (Experimental): One capsule of psilocybin 25 mg will be taken orally with a glass of water.
  Interventions: Drug: Psilocybin 25 mg

INTERVENTIONS:
Drug: Psilocybin 25 mg — The psilocybin used in this study meets quality specifications suitable for human research use. The active drug is encapsulated using a hydroxypropyl methylcellulose (HPMC) capsule and contains 25 mg of psilocybin. The psilocybin will be administered once during the trial in combination with or without risperidone 1 mg. It will also be administered in conjunction with supportive therapy.
  Other Names: PEX010
Drug: Risperidone 1 MG — The risperidone is encapsulated using a cellulose capsule and contains 1 mg of risperidone. The risperidone will be administered once during the trial in combination with psilocybin 25 mg. It will also be administered with supportive therapy.
  Other Names: MAR-Risperidone
  Arms: Risperidone (1 mg) + Psilocybin (25 mg)

SUMMARY:
Limit: 5000 characters. Psilocybin, the chemical component of "magic mushrooms", has been administered with psychotherapy in several randomized clinical trials (RCTs) showing large and sustained antidepressant effects. In healthy volunteers, the psychedelic effects of psilocybin have been shown to be blocked by administration of certain medications such as risperidone.

The purpose of this study is to use an established SV2A radiotracer produced at our Centre to determine the feasibility of integrating PET imaging in to psilocybin trials. The preliminary imaging data will assess whether psilocybin's antidepressant effects are related to changes in synaptic density in adults with TRD, and whether any changes in synaptic density are associated with psilocybin's actions on the 5-HT2AR.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 65 years old;
2. Must be deemed to have capacity to provide informed consent;
3. Must sign and date the informed consent form;
4. Stated willingness to comply with all study procedures;
5. Ability to read and communicate in English, such that their literacy and comprehension is sufficient for understanding the consent form and study questionnaires, as evaluated by study staff obtaining consent;
6. Primary DSM-5 diagnosis of non-psychotic MDD, single or recurrent, based on the Structured Clinical Interview for DSM-5 (SCID-5) administered at the first screening visit;
7. Participants diagnosed with treatment-resistant depression defined as individuals with a baseline HamD-17 score > 14 and that have not responded to two or more separate trials of antidepressants at an adequate dosage and duration (an antidepressant resistance rating score of three or more is considered an adequate trial) based on the Antidepressant Treatment History Form (ATHF); there is no upper limit on the number of treatment failures;
8. Ability to take oral medication;
9. Individuals who are capable of becoming pregnant: use of highly effective contraception for at least 3 months prior to screening and agreement to use such a method during study participation;
10. Individuals who are willing to taper off current antidepressant and antipsychotic medications for a minimum of 2-weeks (or more depending on the medication) prior to Baseline (V2) and whose physician confirms that it is safe for them to do so; and
11. Agreement to adhere to Lifestyle Considerations (section 4.5) throughout study duration.

Exclusion Criteria:

1. Pregnant as assessed by a urine pregnancy test at Screening (V1) or individual's that intend to become pregnant during the study or are breastfeeding;
2. Treatment with another investigational drug or other intervention within 30 days of Screening (V1);
3. Have initiated psychotherapy in the preceding 12 weeks prior to Screening (V1);
4. Have a DSM-5 diagnosis of substance use disorder (use of tobacco is permitted) within the preceding 6 months;
5. Have active suicidal ideation with intent and plan as determined by item 3 of the HamD-17;
6. Any DSM-5 lifetime diagnosis of a schizophrenia-spectrum disorder; obsessive-compulsive disorder, psychotic disorder (unless substance induced or due to a medical condition), bipolar I or II disorder, paranoid personality disorder, borderline personality disorder, or neurocognitive disorder as determined by medical history and the SCID-5 clinical interview;
7. Any first-degree relative with a diagnosis of schizophrenia-spectrum disorder; psychotic disorder (unless substance-induced or due to a medical condition); or bipolar I disorder as determined by the family medical history form and discussions with the participant;
8. Presence of a relative or absolute contraindication to psilocybin, including a drug allergy, recent stroke history, uncontrolled hypertension, low or labile blood pressure, recent myocardial infarction, cardiac arrhythmic, severe coronary artery disease, or moderate to severe renal or hepatic impairment.
9. Presence of baseline prolonged QTc or Torsade de Pointes as measured by the ECG or a history of long QTc syndrome or related risk factors;
10. History of allergy or contraindication to risperidone
11. Current or past traumatic brain injury or other neurological/neurodegenerative disorder
12. Unable or unwilling to undergo PET or MRI scanning (e.g. claustrophobia, pacemaker);
13. Blood disorders, disorders of coagulation, or ongoing use of anticoagulant medication
14. Any disability that may prevent the participant from completing study requirements (e.g., non-correctable clinically significant sensory impairment such as not hearing well enough to communicate with study personnel during scans, or physical disability that does not allow them to lie still on the scanner bed for 1-2 hours);
15. Participant exceeds the annual or lifetime amount of radiation
16. Any other clinically significant physical illness including chronic infectious diseases or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of obtaining PET imaging scans before and after administration of psilocybin (25 mg) with and without risperidone (1 mg). | 24 Months
  Percentage of participants recruited, enrolled, and retained.

SECONDARY OUTCOMES:
Obtain preliminary data on synaptic density (as measured by [18F] SynVesT-1 volume distribution, VT) in brain regions relevant to MDD (i.e., hippocampus, prefrontal cortex) | Before and 4 weeks after administration of psilocybin 25 mg with and without risperidone 1 mg
  as measured by [18F] SynVesT-1 volume distribution, VT

OTHER OUTCOMES:
Change in the Montgomery-Åsberg Depression Rating Scale (MADRS) from Baseline to 1-week post-treatment. | Baseline (Visit 2, Day 0) to 1-week post-treatment (Visit 4, Day 7).
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician-rated scale that measures depression severity. Each item can be scored from 0-6. The minimum assessment score is 0 and the maximum score is 60. Higher composite scores represent a more severe condition.
Obtain preliminary data on cortical plasticity (as measured by TMS-EEG) | Before (visit 2), during (visit 3) and after (visit 4) administration of psilocybin 25 mg with and without risperidone 1 mg
  obtain preliminary data on cortical plasticity, as measured by TMS-EEG in brain regions relevant to MDD at visit 2, visit 3 and visit 4

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ishrat Husain, MBBS, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT06512220/Prot_SAP_001.pdf